CLINICAL TRIAL: NCT06161441
Title: A Phase 2 Peri-Operative Trial of Fianlimab and Cemiplimab in Combination With Chemotherapy Versus Cemiplimab in Combination With Chemotherapy in Patients With Resectable Early Stage (Stage II to IIIB [N2]) NSCLC
Brief Title: A Trial to Learn if the Combination of Fianlimab, Cemiplimab, and Chemotherapy is Safe and Works Better Than the Combination of Cemiplimab and Chemotherapy in Adult Patients With Non-Small Cell Lung Cancer That Can be Treated With Surgery
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R3767-ONC-2266; 2023-505172-29-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Resectable Non-small Cell Lung Cancer
Keywords: Stage II to IIIB (N2); NSCLC; Neoadjuvant therapy; Subsequent adjuvant therapy; PeriOperative
MeSH Terms: interventions — cemiplimab; Pemetrexed; Paclitaxel; Carboplatin; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): Randomized 1:1:1
  Neoadjuvant period:
  placebo + cemiplimab + platinum doublet chemotherapy
  Adjuvant period:
  placebo + cemiplimab
  Interventions: Drug: Cemiplimab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin; Drug: Placebo
- Arm B (Experimental): Randomized 1:1:1
  Neoadjuvant period:
  fianlimab high dose + cemiplimab + platinum doublet chemotherapy
  Adjuvant period:
  fianlimab high dose + cemiplimab
  Interventions: Drug: Fianlimab; Drug: Cemiplimab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin
- Arm C (Experimental): Randomized 1:1:1
  Neoadjuvant period:
  fianlimab low dose + cemiplimab + platinum doublet chemotherapy
  Adjuvant Period:
  fianlimab low dose + cemiplimab
  Interventions: Drug: Fianlimab; Drug: Cemiplimab; Drug: Pemetrexed; Drug: Paclitaxel; Drug: Carboplatin; Drug: Cisplatin

INTERVENTIONS:
Drug: Fianlimab — Administered intravenously (IV) every 3 weeks (Q3W)
  Other Names: REGN3767
  Arms: Arm B; Arm C
Drug: Cemiplimab — Administered IV Q3W
  Other Names: REGN2810; Libtayo
Drug: Pemetrexed — Administered IV Q3W
  Other Names: Alimta
Drug: Paclitaxel — Administered IV Q3W
  Other Names: Taxol
Drug: Carboplatin — Administered IV Q3W
  Other Names: Paraplatin
Drug: Cisplatin — Administered IV Q3W
  Other Names: Platinol
Drug: Placebo — Administered IV Q3W
  Arms: Arm A

SUMMARY:
This study is researching an experimental drug called fianlimab (also called REGN3767) with two other medications called cemiplimab and platinum-doublet chemotherapy, individually called a "study drug" or collectively called "study drugs", when combined in this study. The study is being conducted in patients who have resectable stage II to IIIB (N2) non-small cell lung cancer (NSCLC) that can be treated with surgery.

The aim of the study is to see how effective the combination of fianlimab, cemiplimab, and chemotherapy is in comparison with cemiplimab and chemotherapy as peri-operative therapy in participants with NSCLC.

The study is looking at several other research questions, including:

* What side effects may happen from taking the study drugs
* How much of each study drug is in the blood at different times
* Whether the body makes antibodies against the study drugs (which could make the drugs less effective or could lead to side effects)
* How administering the study drugs might affect quality of life

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients with newly diagnosed, histologically confirmed, fully resectable stage II to IIIB (N2) NSCLC as per American Joint Committee on Cancer (AJCC) version 8
2. For patients with evidence of mediastinal adenopathy on imaging, mediastinal lymph node sampling is required as defined in the protocol
3. All patients must have disease status showing no evidence of distant metastases documented by a complete physical examination and imaging studies performed within 4 weeks prior to randomization as defined in the protocol
4. A patient must have an evaluable Programmed cell death ligand-1 (PD-L1) immunohistochemistry (IHC) result as defined in the protocol
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate bone marrow, hepatic and kidney function as defined in the protocol

Key Exclusion Criteria:

1. Any evidence of locally advanced unresectable or metastatic disease as defined in the protocol
2. Patients with tumors with known Epidermal growth factor receptor (EGFR) gene mutations, anaplastic lymphoma kinase (ALK) gene translocations as defined in the protocol
3. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C virus (HCV) infection as defined in the protocol
4. Treatment with anti-cancer therapy including immunotherapy, chemotherapy, radiotherapy, or biological therapy in the 3 years prior to randomization. Adjuvant hormonotherapy used for breast cancer or other hormone-sensitive cancers in long term remission is allowed.
5. Patients with a history of myocarditis

Note: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-04-17 (Estimated); Study Completion 2029-11-04 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) as evaluated by blinded independent pathological review (BIPR) in post-treatment resected tumor samples | Up to 24 months

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | Up to 3 years
Major pathological response (MPR) by BIPR in post-treatment resected tumor samples | Up to 24 months
MPR by local pathology review in post-treatment resected tumor samples | Up to 24 months
Tumor response to neoadjuvant therapy per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) criteria by investigator assessment | Up to 24 months
Occurrence of Adverse events (AEs) | Up to 5 years
Occurrence of Treatment-emergent adverse event (TEAEs) | Up to 5 years
Occurrence of Serious adverse events (SAEs) | Up to 5 years
Occurrence of Adverse events of special interest (AESIs) | Up to 5 years
Occurrence of immune-mediated adverse events (imAEs) | Up to 5 years
Occurrence of interruption and discontinuation of study drug(s) due to TEAE | Up to 5 years
Occurrence of laboratory abnormalities | Up to 5 years
  Grade ≥3 per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0) including standard hematology, chemistry, urinalysis, and other lab tests
Occurrence of death due to TEAE | Up to 5 years
Concentrations of cemiplimab in serum | Up to 30 months
Concentrations of fianlimab in serum | Up to 30 months
Anti-drug antibodies (ADA) to fianlimab in serum over time | Up to 30 months
ADA to cemiplimab in serum over time | Up to 30 months
Percentage of patients with definitive surgery | Up to 24 months
Percentage of patients with cancelled surgery | Up to 24 months
Percentage of patients with delayed surgery | Up to 24 months
Completeness of resection (R0, R1, R2, Rx) | Up to 24 months
Length in delay of surgery | Up to 24 months
Type of surgery (lobectomy, sleeve lobectomy, bilobectomy, pneumonectomy, other) | Up to 24 months
Median length of hospital stay | Up to 24 months
Surgical approach (thoracotomy, minimally invasive, minimally invasive to thoracotomy) | Up to 24 months
Incidence of peri operative AE associated with surgery | Up to 90 days post-surgery
Incidence of peri operative SAE associated with surgery | Up to 90 days post-surgery
Incidence of post operative AE associated with surgery | Up to 90 days post-surgery
Incidence of post operative SAE associated with surgery | Up to 90 days post-surgery
Overall change in patient-reported global health status/QoL per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Up to 5 years
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Overall change in patient-reported physical functioning per EORTC QLQ-C30 | Up to 5 years
Overall change in patient-reported role functioning per EORTC QLQ-C30 | Up to 5 years
Overall change in patient-reported chest pain per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer 13 (EORTC QLQ-LC13) | Up to 5 years
  The EORTC QLQ-LC13 is a lung cancer-specific supplemental questionnaire used in combination with the EORTC QLQ-C30. Participant responses to the question "Have you had pain in your chest?" are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. The change from baseline in chest pain (EORTC QLQ-LC13 Item 40) score will be presented. A lower score indicates a better outcome.
Overall change in patient-reported dyspnea per EORTC QLQ-LC13 | Up to 5 years
Overall change in patient-reported cough per EORTC QLQ-LC13 | Up to 5 years
Overall change in patient-reported composite of chest pain, dyspnea, and cough per EORTC QLQ-LC13 | Up to 5 years
Change in patient-reported general health status per EuroQoL 5-Dimensional 5-Level Scale (EQ-5D-5L) index | Up to 5 years
  The EQ-5D-5L descriptive system assesses 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a 5-level scale: no problems, slight problems, moderate problems, severe problems and extreme problems
Change in patient-reported general health status per Visual analogue scale (VAS) scores | Up to 5 years
  The EQ-5D-5L VAS records the respondent's self-rated health on a 10 centimeter (cm) vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine".
Time until definitive deterioration in patient-reported global health status/QoL per EORTC QLQ-C30 | Up to 5 years
Time until definitive deterioration in patient-reported physical functioning per EORTC QLQ-C30 | Up to 5 years
Time until definitive deterioration in patient-reported role functioning per EORTC QLQ-C30 | Up to 5 years
Time until definitive deterioration in patient-reported chest pain per EORTC QLQ-LC13 | Up to 5 years
Time until definitive deterioration in patient-reported dyspnea per EORTC QLQ-LC13 | Up to 5 years
Time until definitive deterioration in patient-reported cough per EORTC QLQ-LC13 | Up to 5 years
Time until definitive deterioration in patient-reported composite of chest pain, dyspnea and cough per EORTC QLQ-LC13 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (123):
- United States (8):
  - Clermont Oncology Center, Clermont, Florida
  - University of Illinois, Chicago, Illinois
  - University of Kansas Cancer Center-Westwood, Westwood, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - Mercy South, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - Kaiser Permanente Northwest, Portland, Oregon
  - Virginia Cancer Care Specialist, PC, Fairfax, Virginia
- Australia (3):
  - Eastern Health, Box Hill, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria
  - St John of God Murdoch Hospital, Murdoch, Western Australia
- Chile (4):
  - Orlandi Oncologia, Providencia, Metropolitan Region
  - Clinica Santa Maria, Santiago, Providencia
  - Centro de Oncologia de Precision, Las Condes, Region Metropolitana, Santiago
  - Oncocentro APYS, Viña del Mar, Región de Valparaíso
- France (10):
  - Centre de Oncologie de Gentilly, Nancy, Grand Est
  - Institut de Cancerologie de l'Ouest, Saint-Herblain, Nantes
  - Centre Hospitalier Universitaire (CHU) Bordeaux, Bordeaux, Nouvelle-Aquitaine
  - CHU Limoges, Limoges, Nouvelle-Aquitaine
  - APHP - Hopital Ambroise Pare, Boulogne-Billancourt
  - CHU Dijon, Dijon
  - Centre Hospitalier Universitaire de Nantes Hopital Guillaume et Rene Laennec, Nantes
  - Uneos - Hopital R Schuman, Vantoux
  - Chi Creteil, Créteil, Île-de-France Region
  - Hopital Cochin, Paris, Île-de-France Region
- Georgia (9):
  - Cancer Center of Adjara, Batumi
  - Israeli Georgian Medical Research Clinic Helsicore, Tbilisi
  - Llc Todua Clinic, Tbilisi
  - LTD New Hospitals, Tbilisi
  - High Technology Medical Center, University Clinic Tbilisi, Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - JSC K. Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - TIM - Tbilisi Institute of Medicine, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
- Germany (8):
  - LKI LUngenfachklinik Immenhausen, Immenhausen, Hesse
  - Evang. Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - LungenClinic, Großhansdorf, Schleswig-Holstein
  - Klinikum Esslingen, Esslingen am Neckar
  - Universitatsklinium Giesse, Giessen
  - Asklepios Klinikum Harburg, Hamburg
  - Lungenklinik Hemer, Hemer
  - MVZ fuer Haematologie und Onkologie Rhein-Kreis GmbH, Neuss
- Italy (21):
  - UOC Oncoematologia AOU Vanvitelli, Naples, Campania
  - Istituti di Ricovero e Cura a Carattere Scientifico (IRCCS) Pascale, Napoli, Campania
  - Azienda Ospedaliero-Universitaria Ferrara (AOU Ferrara), Ferrara, Emilia-Romagna
  - AUSL Piacenza, Piacenza, Emilia-Romagna
  - Careggi University Hospital, Florence, Firenze
  - UOC Oncologia Medica Ospedale Civile di Livorno Azienda Usl Toscana Nord Ovest, Livorno, Livorno
  - ASST Ospedale Papa Giovanni XXIII, Bergamo, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milano
  - Azienda Sanitaria Territoriale di Pesaro e Urbino, Pesaro, Pesaro And Urbino
  - Azienda Ospedaliera Nazionale SS Antonio e Biagio e Cesare Arrigo, Alessandria, Piedmont
  - Centro di Riferimento Oncologico (CRO) - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS), Aviano, Pordenone
  - FPO- IRCCS, Istituto di Candiolo, Candiolo, Turin
  - Azienda Ospedaliera Universitaria Pisana, Pisa, Tuscany
  - Istituto Tumori Giovanni Paolo II (Istituto di Ricovero e Cura a Carattere Scientifico Bari), Bari
  - ASST Cremona, Cremona
  - Niguarda Cancer Center, Milan
  - Azienda Ospedaliero-Universitaria Maggiore della Carita - Oncology, Novara
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario Campus Bio-Medico, Roma
  - Instituto Fisioterapici Ospitalieri (IFO) Istituto Regina Elena, Rome
  - Azienda Sanitaria Universitaria Friuli Centrale (ASU FC) Santa Maria della Misericordia, Udine
- Malaysia (4):
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur, Negeri / Wilayah Persekutuan
  - Hospital Pulau Pinang, George Town, Pulau Pinang
  - Hospital Umum Sarawak, Kuching
- South Korea (9):
  - National Cancer Center, Gyeonggi-do, Gyeonggi-do
  - The Catholic University of Korea St Vincents Hospital, Suwon, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Gachon University Gil Medical Center, Incheon, Namdong-Gu
  - Inha University Hospital, Incheon
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (19):
  - Hospital Clinico Universitario Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital General Universitario Elche, Elche, Alicante
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Son Espases, Palma, Balearic Islands
  - IOB Institute of Oncology Quiron, Barcelona, Catalonia
  - Instituto Oncologico Dr Rosell, Barcelona, Catalonia
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - Alvaro Cunqueiro Hospital, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Althaia - Xarxa Assistencial Universitaria de Manresa - Orde Hospitalaria de Sant Joan de Deu, Barcelona
  - Catalan Institute of Oncology, Girona
  - Hospital Universitario Lucus Augusti, Lugo
  - Fundacion Jimenez Diaz, Madrid
  - Hospital 12 de Octubre, Madrid
  - Hospital De Valme, Seville
  - Fundacion IVO, Valencia
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia
- Taiwan (9):
  - Changhua Christian Hospital, Changhua, Changhua County
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin
  - Hualien Tzu Chi Hospital, Hualien City
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wan Fang Hospital, Taipei
- Turkey (Türkiye) (19):
  - Acibadem Adana Hastanesi, Adana, Adana
  - Ege University Faculty of Medicine, Bornova, İzmir
  - Kocaeli University Hospital, Kocaeli, Marmara
  - Faculty of Medicine of Sakarya University, Sakarya, Marmara
  - Necmettin Erbakan University Meram Faculty of Medicine, Konya, Meram
  - Ondokuz Mayıs University, Kurupelit, Samsun
  - Medical Point Gaziantep Hastanesi, Gaziantep, Sehitkamil
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Yenimahalle
  - Baskent University Adana Turgut Noyan Hospital, Adana, Yuregir
  - Adana City Education and Research Hospital, Adana, Yuregir
  - Gulhane Training and Research Hospital, Ankara
  - Liv Hospital Ankara, Ankara
  - Hacettepe University Cancer Institute, Ankara
  - Memorial Ankara Hospital, Ankara
  - Ankara University Faculty of Medicine, Ankara
  - Koc University, Istanbul
  - Bezmialem Vakif University, Istanbul
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Istanbul Medeniyet University Prof.Dr.Suleyman Yalcin Şehir Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/